CLINICAL TRIAL: NCT06533020
Title: Long-term Outcomes of Complex Conversion Total Hip Arthroplasty
Acronym: LOCC
Status: Active, not recruiting | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Other Study IDs: 24-1026
Record Dates: First submitted 2024-07-24; First posted 2024-08-01 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Arthroplasty Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Complex Total Hip Arthroplasty: Participants who have undergone complex total hip arthroplasty within the last 10 years
- Conversion Total Hip Arthroplasty: Participants who have undergone conversion total hip arthroplasty within the last 5 years

SUMMARY:
The purpose of the research study is to examine the long-term outcomes of complex and conversion total hip arthroplasty procedures. By means of both retrospective (chart review) and prospective (in-person clinic visits) radiographs and validated patient-reported outcome scores including the Hip Disability and Osteoarthritis Outcome Score (HOOS) and the Patient-Reported Outcomes Measurement Information System (PROMIS), the research team aims to collect, analyze, and summarize the outcome data. The outcomes of the follow-up appointment will be analyzed in comparison to previous findings over various intervals to assess changes over time, if data is available.

ELIGIBILITY:
Inclusion Criteria:

* Having undergone a conversion total hip arthroplasty (THA) more than five years ago or a complex THA more than ten years ago done by a UNC Health-affiliated physician
* Willingness to receive follow-up care from a UNC Health-affiliated physician or provide outcome data regarding this surgical intervention
* Able to speak and read English
* Able to consent to participation

Exclusion Criteria:

* Less than 18 years of age
* Incarcerated status

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: UNC Orthopaedics
Sampling Method: Non-Probability Sample
Enrollment: 210 (Estimated)
Dates: Start 2024-10-06 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
PROMIS SF v1.1-Pain Interference 8a | once during the 36-month total study duration, preferably during initial recruitment, but open to collection at any time during the study timeframe
  The Patient-Reported Outcomes Measurement Information System (PROMIS) SF v1.1-Pain Interference 8a measures the amount of pain interference in daily life. Possible scores range from "not at all" (1) to "very much" (5), with higher scores indicating a worse outcome (more pain interference).
PROMIS SF v2.0 - Physical Function 20a | once during the 36-month total study duration, preferably during initial recruitment, but open to collection at any time during the study timeframe
  The Patient-Reported Outcomes Measurement Information System (PROMIS) SF v2.0 - Physical Function 20a measures the level of individual physical function in daily life. Possible scores range from "without any difficulty" (1) to "unable to do" (5) and "not at all" (1) to "cannot do" (5), with higher scores indicating a worse outcome (less physical function ability).
HOOS | once during the 36-month total study duration, preferably during initial recruitment, but open to collection at any time during the study timeframe
  The Hip Disability and Osteoarthritis Outcome Score (HOOS) measures an individual's feelings about their hip and how well they are able to do usual activities, based on symptoms, stiffness, pain, daily living function, sports and recreational activities function, and quality of life. Possible scores range from "never" (1) to "always" (5) and "none" (1) to "extreme" (5), with higher scores indicating a worse outcome.
Radiographic Findings | once during the 36-month total study duration, preferably during screening for initial recruitment, but open to collection at any time during the study timeframe
  Standard radiographs of implanted hip to assess device efficacy and other potential anomalies. Collected during in-person clinic visits or from chart review if the patients have had hip radiographs at UNC in the past two years.

SECONDARY OUTCOMES:
Number of participants with comorbidities | Up to 36-months total study duration
  Individual health statuses (as diagnosed and present in the electronic medical record (EMR) throughout patient lifespan) thought to complicate the surgical procedure and recovery. Retrospectively collected during chart review including 20 statuses such as Diabetes Mellitus, Autoimmune Disorders, Current Immunosuppression, Current Dialysis/End Stage Renal Disease (ESRD), Chronic Kidney Disease (I-III), Heart Failure, Coronary Artery Disease, etc.
Number of participants with complications | Up to 36 months total study duration
  Individual health events (as present in the EMR throughout patient lifespan) and risk factors complicating the surgical procedure and recovery. Retrospectively collected during chart review including several events such as Iatrogenic fracture, Bleeding (Blood Transfusion), Surgical Site Infection, THA Periprosthetic Fracture, Wound Complication, etc, and risk factors such as Hip surgery prior to THA, age > 70, Drug/alcohol use, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Alecia Rajesh, Principal Investigator — University of North Carolina, Chapel Hill; Ishani Deliwala, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Supporting Information: Study Protocol, ICF
Time Frame: Beginning 9 and continuing 36 months following publication
Access Criteria: Investigator has approved IRB, IEC REB and an executed data use/sharing agreement with UNC.